CLINICAL TRIAL: NCT01602757
Title: An Open-Label Pharmacokinetic Study of the Synera Patch Applied for 2-, 4-, and 12-hours and a Lidocaine/Tetracaine Patch Without Heat Applied for 4 Hours in Healthy Adult Volunteers
Brief Title: Pharmacokinetic Study of Synera in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SC-101
Record Dates: First submitted 2012-05-15; First posted 2012-05-21 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine; Tetracaine; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synera (Experimental): Subjects received 4 Synera® patches for 2 hours in Session 1 and 4 patches for 12 hours in Session 4. During Study Session 2, subjects were randomly assigned to 4-hour applications of either 4 Synera® patches or 4 lidocaine/tetracaine patches without heat ("no heat patches") and were crossed over during Study Session 3.
  Interventions: Drug: Synera

INTERVENTIONS:
Drug: Synera — Subjects received 4 Synera® patches for 2 hours in Session 1 and 4 patches for 12 hours in Session 4. During Study Session 2, subjects were randomly assigned to 4-hour applications of either 4 Synera® patches or 4 lidocaine/tetracaine patches without heat ("no heat patches") and were crossed over during Study Session 3.
  Other Names: Lidocaine 70 mg/Tetracaine 70 mg topical patch

SUMMARY:
This study will measure the amount of lidocaine and tetracaine in the blood after 2-, 4-, and 12-hour application of 4 Synera patches and a 4 hour application of 4 patches without heat.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the pharmacokinetic profiles of lidocaine and tetracaine after 2-, 4-, and 12-hour application of 4 Synera® patches and a 4-hour application of 4 lidocaine/tetracaine patches without heat in healthy adult subjects and to monitor the frequency and nature of adverse events. In addition to determining the pharmacokinetics for a one-time application of 4 Synera® patches, steady-state pharmacokinetics were modeled and residual patch concentrations of lidocaine and tetracaine were determined.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* be a nonsmoker
* have a body mass index (BMI) ≥ 18.5 and < 30.0

Exclusion Criteria:

* known or suspected hypersensitivity, allergies, or other contraindications to any compound present in the study drug, including lidocaine, tetracaine, or other local anesthetics.
* have a defect, injury or a dermatological disease or condition in the skin area where the study drug was to be applied.
* have a history or current evidence of any hepatic impairment.
* have failed the urine drug screen.
* have used or been administered a local or systemic anesthetic, including over-the-counter products, within the past 14 days.
* have donated blood or plasma within the past 30 days.
* have participated in a clinical research study within the past 30 days.
* are pregnant, breastfeeding, or was a female of childbearing potential and not practicing adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of Synera after application of 4 patches | 0.5, 1, 1.5, 2, 4, 8, 10, 12 hours post-dose
  Peak plasma concentration of Synera after application of 4 patches for 2-, 4- and 12-hours

SECONDARY OUTCOMES:
Number of participants with adverse events | 24 days
Area under the plasma concentration versus time (AUC) of Synera | 0.5, 1, 1.5, 2, 4, 8, 10, 12 hours post-dose
  Area under the plasma concentration versus time curve of Synera after application of 4 patches for 2-, 4-, and 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Result] Marriott TB, Charney MR, Stanworth S. Effects of application durations and heat on the pharmacokinetic properties of drug delivered by a lidocaine/tetracaine patch: a randomized, open-label, controlled study in healthy volunteers. Clin Ther. 2012 Oct;34(10):2174-83. doi: 10.1016/j.clinthera.2012.08.008. Epub 2012 Sep 1. PMID 22943969